CLINICAL TRIAL: NCT04566250
Title: Non-Opioid Prescriptions After Arthroscopic Surgery in Canada (NO PAin): a Randomized Controlled Trial
Brief Title: Non-Opioid Prescriptions After Arthroscopic Surgery in Canada (NO PAin)
Acronym: NO PAin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Olufemi Ayeni, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NOPain1111
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Knee Arthroscopy; Shoulder Arthroscopy

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized using the centralized 24-hour computerized randomization system to allocate patients to the control (standard of care) or intervention (non-opioid prescription and infographic) group.
Who Masked: Outcomes Assessor
Masking Description: Given that patients in the intervention group will receive a pamphlet explaining how to use their prescription allocation, patient blinding is not feasible. Surgeons cannot be blinded as they will need to sign the prescriptions and provide any necessary advice about the medications being prescribed. Outcome assessors and data analysts will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-Opioid Prescription and Infographic (Active Comparator): The study intervention will involve 3 components:
  1. A standardized non-opioid prescription: A prescription for Naproxen 500mg PO BID PRN x 60 tabs, Acetaminophen 1000mg PO Q6H PRN x 100 500mg tabs and Pantoprazole 20mg PO daily x 30 tabs (to be taken only while utilizing Naproxen). In the case of a Naproxen intolerance, a prescription for Meloxicam 15mg PO BID PRN x 60 tabs will be given.
  2. A limited opioid "rescue prescription": A prescription of Hydromorphone 1mg PO Q4H PRN x 10 tabs will be included on a separate prescription.
  3. Patient education infographic: The infographic will contain information on how to take the prescribed medications, along with instructions that the morphine rescue prescription should only be used in cases where the non-opioid pain medications are not providing satisfactory pain control.
  Interventions: Combination Product: Non-Opioid Prescription and Infographic
- Standard of Care (Other): The control group is standard of care, which typically includes a prescription for an opioid.
  Interventions: Combination Product: Non-Opioid Prescription and Infographic

INTERVENTIONS:
Combination Product: Non-Opioid Prescription and Infographic — The study intervention will involve 3 components:
  1. A standardized non-opioid prescription: A prescription for Naproxen 500mg PO BID PRN x 60 tabs, Acetaminophen 1000mg PO Q6H PRN x 100 500mg tabs and Pantoprazole 40mg PO daily x 30 tabs (to be taken only while utilizing Naproxen).
  2. A limited opioid "rescue prescription": A prescription of Hydromorphone 1mg PO Q4H PRN x 10 tabs will be included on a separate prescription.
  3. Patient education infographic: The infographic will contain information on how to take the prescribed medications, along with instructions that the morphine rescue prescription should only be used in cases where the non-opioid pain medications are not providing satisfactory pain control.

SUMMARY:
This is a randomized controlled trial of 200 patients between the ages of 18 and 65 years undergoing outpatient knee or shoulder arthroscopy. Patients will be evaluated clinically at 2 and 6 weeks post-operatively. Patients will be recruited from experienced arthroscopic surgeons at 3 hospital sites in Hamilton, Ontario. All research will be conducted according to international standards of Good Clinical Practice and institutional research policies and procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing outpatient knee or shoulder arthroscopy for any of the following procedures: ACL reconstruction (with or without LET), MPFL reconstruction (not including TTO), Chondroplasty, Meniscectomy, Meniscal repair Meniscal transplant, Microfracture, ACI, Fixation of unstable osteochondral lesion, Subacromial decompression, Rotator cuff repair, Shoulder stabilization, Superior capsule reconstruction, Biceps tenotomy/tenodesis, Capsular release, SLAP repair, Diagnostic arthroscopy, Irrigation and/or debridement, Loose body removal, Synovectomy
2. Patients aged 18 years and older
3. Patients who have the ability to speak, understand, and read English
4. Provision of informed consent

Exclusion Criteria:

1. Patients who take or are on a home dose of an opioid medication (i.e. once daily or more)
2. Patients involved in ongoing litigation or compensation claims for any injury (e.g. Work Safety Insurance Board, WSIB)
3. Patients involved in another research study that requires a specific post-operative pain control medication regimen
4. Patients undergoing a knee or shoulder arthroscopy procedure that will likely have an operative time greater than 3 hours
5. Patients who will undergo concomitant open surgery
6. Patients who require overnight admission
7. Patients with a contraindication or allergy to NSAIDs, acetaminophen, or morphine and hydromorphone
8. Patients diagnosed with renal disease or cardiac disease
9. Patients who are scheduled for/plan to have an additional surgical procedure during the 6-week follow-up period
10. Patients who will likely have problems, in the judgement of the investigator, with maintaining follow-up
11. Any other reason(s) the investigator feels is relevant for excluding the patient

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Total oral morphine equivalents (OMEs) | 6 weeks postoperatively
  The primary outcome is the number of total OMEs consumed as determined by a patient-reported medication diary.

SECONDARY OUTCOMES:
Pain (Visual Analogue Scale, VAS) | 6 weeks postoperatively
  The VAS will include a 100mm line, on which patients will be asked to rate their average pain since their surgery.
Patient Satisfaction (Hospital Consumer Assessment of Health Care Provider and Systems Question, HCAHPS) | 6 weeks postoperatively
  We used the following modified question from the HCAHPS questionnaire related to satisfaction with pain relief, answered on a Likert scale (never, sometimes, usually, or always): "In the time after surgery, how often was your pain well controlled?"
OMEs Prescribed | 6 weeks postoperatively
  As per the medication diary
Opioid Refills | 6 weeks postoperatively
  As per the medication diary
Adverse Events | 6 weeks postoperatively
  Adverse events, defined as any symptom, sign, illness, or experience that develops or worsens in severity during the course of this study, will be documented.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Hamilton General Hospital, Hamilton, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No
No data sharing

REFERENCES:
- [Derived] NO PAin Investigators; Gazendam A, Ekhtiari S, Horner NS, Simunovic N, Khan M, de Sa DL, Madden K, Ayeni OR. Effect of a Postoperative Multimodal Opioid-Sparing Protocol vs Standard Opioid Prescribing on Postoperative Opioid Consumption After Knee or Shoulder Arthroscopy: A Randomized Clinical Trial. JAMA. 2022 Oct 4;328(13):1326-1335. doi: 10.1001/jama.2022.16844. PMID 36194219
- [Derived] NO PAin Investigators. Protocol for a multicenter randomized controlled trial comparing a non-opioid prescription to the standard of care for pain control following arthroscopic knee and shoulder surgery. BMC Musculoskelet Disord. 2021 May 22;22(1):471. doi: 10.1186/s12891-021-04354-x. PMID 34022863